CLINICAL TRIAL: NCT00566488
Title: Parathyroid and Thymus Transplantation in DiGeorge Syndrome, #931
Brief Title: Parathyroid and Thymus Transplantation in DiGeorge #931
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma Switzerland GmbH (Industry)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency); National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00016482; R01AI047040 (NIH); 5K12HD043494-09 (NIH); R01AI054843 (NIH); FDA-FD-R-002606 (Other Grant/Funding Number: FDA); 2R01AI047040-11A2 (NIH); R56 Bridge R01AI4704011A1 (Other Grant/Funding Number: [NIH American Recovery and Reinvestment Act (ARRA) of 2009]); 3R56AI047040-11A1S1 (NIH); #931
Record Dates: First submitted 2007-11-30; First posted 2007-12-03 (Estimated); Last update posted 2022-04-04 (Actual); Status verified 2020-04

CONDITIONS: DiGeorge Syndrome; Hypoparathyroidism; Complete DiGeorge Syndrome
Keywords: Thymus Transplantation; Parathyroid Transplantation; DiGeorge Syndrome; Hypoparathyroidism; Athymia
MeSH Terms: conditions — DiGeorge Syndrome; Hypoparathyroidism; Thymic aplasia | interventions — Thymus Extracts

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Thymus and Parathyroid transplantation (Experimental): Thymus/Parathyroid Transplantation in Complete DiGeorge Syndrome Infants
  Interventions: Biological: Thymus/Parathyroid Transplantation

INTERVENTIONS:
Biological: Thymus/Parathyroid Transplantation — Thymus tissue, thymus donor, mother of thymus donor, & parental parathyroid donor screened for transplant safety. Depending on T cell phenotype & function, subjects were given 1 of 2 immunosuppression regimes. All received rabbit anti thymocyte globulin pretransplantation. Others also received cyclosporine pre & post-transplantation. The thymus dose was over 0.2 grams/kg recipient weight. Thymus transplant occurred in operating room; thymic slices were placed in quadriceps. Parathyroid harvest was done under general anesthesia. One parathyroid gland was minced and placed in quadriceps muscle. There was no dose in mg. An open biopsy of thymus allograft was done 2-3 months post-transplant. Biopsy tissue was examined by immunohistochemistry to evaluate for thymopoiesis & graft rejection.
  Other Names: IND 9836, Thymus Tissue

SUMMARY:
This study has three primary purposes: to assess parathyroid function after parathyroid transplantation in infants with Complete DiGeorge syndrome; to assess immune function development after transplantation; and, to assess safety and tolerability of the procedures. This is a Phase 1, single site, open, non-randomized clinical protocol. Enrollment is closed and study intervention is complete for all enrolled subjects; but subjects continue for observation and follow-up. Subjects under 2 years old with complete DiGeorge syndrome (atypical or typical) received thymus transplantation. Subjects received pre-transplant immune suppression with rabbit anti-human-thymocyte-globulin. Subjects with hypoparathyroidism and an eligible parental donor received thymus and parental parathyroid transplantation. A primary hypothesis: Thymus/Parathyroid transplant subjects will need less calcium and/or calcitriol supplementation at 1 year post-transplant as compared to historical controls.

DETAILED DESCRIPTION:
Detailed: DiGeorge Syndrome is a complex of three problems, 1) cardiac defects, 2) parathyroid deficiency, and 3) absence of the thymus, resulting in profound T-cell deficiency. There is a spectrum of disease in DiGeorge syndrome with respect to all three defects. There is no safe and effective treatment for DiGeorge Syndrome and most patients die by the age of two. For patients with a severe T cell defect, the PI has shown that thymus transplantation is safe and efficacious under other clinical protocols. Subjects with complete typical and atypical DiGeorge syndrome were eligible for this study. Subjects with athymia and profound hypoparathyroidism were eligible for parental parathyroid transplantation in this protocol. DiGeorge syndrome infants, who have successful thymus transplants but have hypoparathyroidism, must go to the clinic for frequent calcium levels and to the hospital for calcium infusions; infants with hypoparathyroidism are at risk for seizures from low calcium. Approximately ½ of infants with profound hypoparathyroidism will develop nephrocalcinosis. Depending on T cell phenotype and function, subjects were given one of two different immunosuppression regimens. Typical complete DiGeorge subjects (with proliferative T cell function < 50,000 cpm) received Thymoglobulin pre-transplantation. Typical complete DiGeorge subjects (with proliferative cell response to PHA > 50,000 cpm) and atypical DiGeorge subjects (with proliferative T cell response to PHA < 75,000 cpm) received Thymoglobulin (pre-transplantation) and cyclosporine (pre-transplantation and post-transplantation). Thymoglobulin was used in part to prevent graft rejection and also to deplete any T cells in the donor parathyroid. Cyclosporine was used to deplete activated T cells in the recipient. For all subjects, acetaminophen, diphenhydramine, and methylprednisolone were given concurrently with the rabbit anti-human thymocyte globulin. The thymus was cultured in standard medium for 10-21 days to deplete mature thymocytes which could cause GVHD. In the operating room, thymus tissue was placed in the quadriceps muscle in one or both legs. The parathyroid donation was preferably done at the same time as the thymus transplantation. Parathyroid tissue was placed in the quadriceps muscle in only one leg, using the same incision as the thymus transplantation. Depending on post-transplant immune status, subjects may have received cyclosporine and steroids.

For 3 months after thymus transplantation, T cells were monitored by flow cytometry approximately every 2-4 weeks. Alternatively, absolute lymphocyte count was used as the maximum possible T cell number. At 2-3 months post-transplant, the subject may have had a thymus allograft biopsy, done under general anesthesia in the operating room. The biopsy was approximately 4 pea-sized (3x3mm) portions of muscle tissue where the thymus transplant had been inserted. Using immunohistochemistry, the biopsy determined thymopoiesis and any graft rejection. The parathyroid was not biopsied because it is very small; doing a biopsy could remove all of the parathyroid tissue. A research skin biopsy (at site of skin incision at the time of transplantation) was done to determine whether T cells were present pre-transplantation. A skin biopsy was also done at the time of thymus graft biopsy to look for clonal T cell populations. For all subjects who developed T cells, post-transplantation pneumocystis prophylaxis was used for approximately 1 year and IV immunoglobulin for approximately 2 years.

ELIGIBILITY:
Transplant Inclusion:

* Complete DiGeorge syndrome (typical or atypical) - may have DiGeorge as part of 22q11 hemizygosity, CHARGE association, or diabetic embryopathy or they may have no associated syndromes.
* Must have 1 of following:

  * Circulating CD3+ T cells < 50/mm3; or
  * Circulating CD3+ T cells that also positive for CD45RA and CD62L must be <50/mm3 or must be < 5% of total T cells.
* Must be <24 months old
* Laboratory studies must be done w/in 1 month of treatment:

  * Thyroid studies - if abnormal must be on therapy, if recommended by endocrinology:
  * PT and PTT must be <2x upper limits of normal (ULN)
  * Absolute neutrophil count must be >500/mm3
  * Platelet count must be >50,000/mm3
  * AST and ALT must be <5x ULN
  * Creatinine must be <1.5 mg/dl
* Parents must agree to have infant stay in Durham until thymus biopsy is done 2-3 months post-treatment.
* Typical subjects must not have a rash with T cells on biopsy nor lymphadenopathy.
* Atypical subjects have rash with T cells on biopsy; may have lymphadenopathy.
* PHA proliferative responses must be tested 2x • Atypical: PHA response must be <75,000cpm on 2 tests; test can be done while on immunosuppression.

Additional Criteria for Parathyroid Treatment Inclusion

* Hypoparathyroidism
* At least 1 parent must agree to be parathyroid donor
* Must require calcium supplementation to maintain ionized calcium >1.0 mmol/L. Alternatively, intact PTH must be <lower limit of normal when ionized calcium is <1.2 mmol/L. (Intact PTH measured 2x pre-treatment.)

DiGeorge Treatment Exclusion:

* Heart surgery conducted <4 weeks pre-treatment
* Heart surgery anticipated w/in 3 months of treatment
* Rejection by surgeon or anesthesiologist as surgical candidate
* Lack of sufficient muscle tissue to accept 0.2gms/kg treatment
* Prior attempts at immune reconstitution, such as bone marrow treatment or previous thymus treatment
* Doesn't commit to remaining at Duke until thymus allograft biopsy

Parathyroid Donor Inclusion:

* Serum calcium in normal range
* Normal parathyroid hormone function
* HLA typing must be consistent with parentage.
* Must not be on anticoagulation or can come off
* Parent chosen for donation will be the 1 sharing most HLA alleles with thymus donor
* HLA-DR matching preferred over HLA class I matching. If there no HLA matching at all, then either parent will be acceptable if meets other criteria.
* Negative for EBV; CMV; HIV-1; Syphilis; West Nile virus; Hepatitis B; Hepatitis C; pregnancy; & evidence of head/neck infection
* Fiberoptic nasolaryngoscopy shows vocal cords functioning normally.
* Normal thyroid function
* No history of cancer
* The infant-recipient has 2 living involved parents.

Parathyroid Donor Exclusion:

* Infant recipient doesn't have 2 living involved parents
* Animal tissue/organ recipient
* EBV
* CMV
* HIV-1
* Syphilis
* West Nile virus
* Hepatitis B
* Hepatitis C
* Pregnant
* Evidence of head/neck infection
* Vocal cords not functioning normally.
* Thyroid abnormalities
* Hyperparathyroidism
* History of cancer
* Mad cow disease (positive)
* SARS(and exposure)
* Smallpox exposure

Biological Mother of DiGeorge Subjects Inclusions:

Mother must be competent to consent or assent to study participation and willing to provide blood sample. No other inclusion/exclusion.

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2005-01; Primary Completion 2007-08 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Efficacy parameter: use of calcium/calcitriol at 1 year post-transplantation. | 1 year after thymus transplantation
  Subjects wtih complete DiGeorge anomaly who have received thymus and parathyroid transplants and survived to one year

SECONDARY OUTCOMES:
Efficacy parameters: ionized calcium | 10-14 months after thymus transplantation
  Ionized calcium (normal values are 1.2 - 1.37 mmol/L)
Efficacy parameters: CD3 count | 10-14 months after thymus transplantation
  CD3 count/mm3
Efficacy parameters: CD4 count | 10-14 months after thymus transplantation
  CD4 count/mm3
Efficacy parameters: CD8 count | 10-14 months after thymus transplantation
  CD8 count/mm3
Efficacy parameters: naive CD4 count | 10-14 months after thymus transplantation
  naive CD4 count/mm3
Efficacy parameters: naive CD8 count | 10-14 months after thymus transplantation
  naive CD8 count/mm3
Efficacy parameters: proliferative response to phytohemagglutinin | approximately 1 year after thymus transplantation (8.9 to 17.8 months after transplantation)
  proliferative response to phytohemagglutinin in counts per minute
Efficacy parameters: proliferative response to tetanus toxoid | approximately 1 year after thymus transplantation (8.9 to 17.8 months after transplantation)
  proliferative response to tetanus toxoid in counts per minute
Efficacy parameters: spectra typing at 1 year post transplantation | approximately 1 year after thymus transplantation (12.1 to 18.0 months after transplantation)
  Variability of CD4 T cell receptor beta repertoire as assessed by the Kullback-Leibler divergence (DKL)

CONTACTS AND LOCATIONS:
Overall Officials: M. Louise Markert, MD, PhD, Principal Investigator — Duke University Medical Center, Pediatrics, Allergy & Immunology
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Markert ML, Marques JG, Neven B, Devlin BH, McCarthy EA, Chinn IK, Albuquerque AS, Silva SL, Pignata C, de Saint Basile G, Victorino RM, Picard C, Debre M, Mahlaoui N, Fischer A, Sousa AE. First use of thymus transplantation therapy for FOXN1 deficiency (nude/SCID): a report of 2 cases. Blood. 2011 Jan 13;117(2):688-96. doi: 10.1182/blood-2010-06-292490. Epub 2010 Oct 26. PMID 20978268
- [Background] Chinn IK, Devlin BH, Li YJ, Markert ML. Long-term tolerance to allogeneic thymus transplants in complete DiGeorge anomaly. Clin Immunol. 2008 Mar;126(3):277-81. doi: 10.1016/j.clim.2007.11.009. Epub 2007 Dec 26. PMID 18155964
- [Background] Selim MA, Markert ML, Burchette JL, Herman CM, Turner JW. The cutaneous manifestations of atypical complete DiGeorge syndrome: a histopathologic and immunohistochemical study. J Cutan Pathol. 2008 Apr;35(4):380-5. doi: 10.1111/j.1600-0560.2007.00816.x. PMID 18333898
- [Background] Markert ML, Sarzotti M, Ozaki DA, Sempowski GD, Rhein ME, Hale LP, Le Deist F, Alexieff MJ, Li J, Hauser ER, Haynes BF, Rice HE, Skinner MA, Mahaffey SM, Jaggers J, Stein LD, Mill MR. Thymus transplantation in complete DiGeorge syndrome: immunologic and safety evaluations in 12 patients. Blood. 2003 Aug 1;102(3):1121-30. doi: 10.1182/blood-2002-08-2545. Epub 2003 Apr 17. PMID 12702512
- [Background] Chinn IK, Olson JA, Skinner MA, McCarthy EA, Gupton SE, Chen DF, Bonilla FA, Roberts RL, Kanariou MG, Devlin BH, Markert ML. Mechanisms of tolerance to parental parathyroid tissue when combined with human allogeneic thymus transplantation. J Allergy Clin Immunol. 2010 Oct;126(4):814-820.e8. doi: 10.1016/j.jaci.2010.07.016. Epub 2010 Sep 15. PMID 20832849
- [Background] Chinn IK, Milner JD, Scheinberg P, Douek DC, Markert ML. Thymus transplantation restores the repertoires of forkhead box protein 3 (FoxP3)+ and FoxP3- T cells in complete DiGeorge anomaly. Clin Exp Immunol. 2013 Jul;173(1):140-9. doi: 10.1111/cei.12088. PMID 23607606
- [Result] Markert ML, Devlin BH, Chinn IK, McCarthy EA. Thymus transplantation in complete DiGeorge anomaly. Immunol Res. 2009;44(1-3):61-70. doi: 10.1007/s12026-008-8082-5. PMID 19066739
- [Result] Markert ML, Devlin BH, McCarthy EA, Chinn IK, Hale LP. Thymus Transplantation in Thymus Gland Pathology: Clinical, Diagnostic, and Therapeutic Features. Eds Lavinin C, Moran CA, Morandi U, Schoenhuber R. Springer-Verlag Italia, Milan, 2008, pp 255-267.
- [Result] Markert ML, Devlin BH, Chinn IK, McCarthy EA, Li YJ. Factors affecting success of thymus transplantation for complete DiGeorge anomaly. Am J Transplant. 2008 Aug;8(8):1729-36. doi: 10.1111/j.1600-6143.2008.02301.x. Epub 2008 Jun 28. PMID 18557726
- [Result] Hudson LL, Louise Markert M, Devlin BH, Haynes BF, Sempowski GD. Human T cell reconstitution in DiGeorge syndrome and HIV-1 infection. Semin Immunol. 2007 Oct;19(5):297-309. doi: 10.1016/j.smim.2007.10.002. Epub 2007 Nov 26. PMID 18035553
- [Result] Markert ML, Li J, Devlin BH, Hoehner JC, Rice HE, Skinner MA, Li YJ, Hale LP. Use of allograft biopsies to assess thymopoiesis after thymus transplantation. J Immunol. 2008 May 1;180(9):6354-64. doi: 10.4049/jimmunol.180.9.6354. PMID 18424759
- [Result] Markert ML, Devlin BH, Alexieff MJ, Li J, McCarthy EA, Gupton SE, Chinn IK, Hale LP, Kepler TB, He M, Sarzotti M, Skinner MA, Rice HE, Hoehner JC. Review of 54 patients with complete DiGeorge anomaly enrolled in protocols for thymus transplantation: outcome of 44 consecutive transplants. Blood. 2007 May 15;109(10):4539-47. doi: 10.1182/blood-2006-10-048652. Epub 2007 Feb 6. PMID 17284531
- [Result] Markert ML and Devlin BH. Thymic reconstitution (in Rich RR, Shearer WT, Fleischer T, Schroeder HW, Weyand CM, Frew A, eds., Clinical Immunology 3rd edn., Elsevier, Edinburgh) p 1253-1262, 2008.
- [Result] Markert ML, Devlin BH, McCarthy EA. Thymus transplantation. Clin Immunol. 2010 May;135(2):236-46. doi: 10.1016/j.clim.2010.02.007. Epub 2010 Mar 16. PMID 20236866
- [Result] Markert ML, Alexieff MJ, Li J, Sarzotti M, Ozaki DA, Devlin BH, Sedlak DA, Sempowski GD, Hale LP, Rice HE, Mahaffey SM, Skinner MA. Postnatal thymus transplantation with immunosuppression as treatment for DiGeorge syndrome. Blood. 2004 Oct 15;104(8):2574-81. doi: 10.1182/blood-2003-08-2984. Epub 2004 Apr 20. PMID 15100156